CLINICAL TRIAL: NCT05083351
Title: Performance of Masimo MightySat Pulse Oximeter in Differing Levels of Skin Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1004
Record Dates: First submitted 2021-10-07; First posted 2021-10-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MightySat (Experimental): All subjects who are enrolled into the test group and participate in data collection have the noninvasive MightySat pulse oximeter applied on their finger(s).
  Interventions: Device: MightySat

INTERVENTIONS:
Device: MightySat — Noninvasive pulse oximeter

SUMMARY:
Evaluation of the noninvasive oxygen saturation (SpO2) performance of the noninvasive Masimo MightySat against reference arterial blood samples analyzed by a laboratory CO-oximeter reference instrument. The study will include different subgroups to assess the performance across different genders and skin pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Subject has a hemoglobin value ≥ 11 g/dL.
* Subject's baseline heart rate is ≥ 45 bpm and ≤ 85 bpm.
* Subject's CO value is ≤ 2.0% FCOHb.
* Subject's blood pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* Subject is able to read and communicate in English and understands the study and the risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject has a BMI > 35.
* Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation.*
* Subject has known drug or alcohol abuse.
* Subject uses recreational drugs.*
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
* Subject has any chronic bleeding disorder (e.g. hemophilia).
* Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has any symptomatic cardiac dysrhythmia (e.g. atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (e.g. schizophrenia, bipolar disorder, multiple sclerosis, Huntington's disease) that interferes with the subject's level of consciousness.*
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any active signs and/or symptoms of infectious disease (e.g. hepatitis, HIV, tuberculosis, flu, malaria, measles, etc.).*
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery.*
* Subject has symptoms of congestion, head cold, or other illnesses.
* Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer).*
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to lidocaine, chlorhexidine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes, or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the past 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (working out, riding a bike, riding a skateboard, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MightySat
Started | 88
Completed | 39
Not Completed | 49
Not completed — Adverse Event | 3
Not completed — Did not meet data inclusion criteria | 8
Not completed — Did not meet eligibility criteria | 19
Not completed — Study Staff Decision | 19

BASELINE CHARACTERISTICS:
Arm/Group | MightySat
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 9
  More than one race | 5
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Accuracy of the MightySat Pulse Oximeter
Description: The SpO2 accuracy of the MightySat pulse oximeter was determined by calculating the root mean-squared (rms) difference between the measured values (SpO2) to the reference values (SaO2) in accordance with ISO-80601-2-61.
  Arms= √(∑(i=1 to n) ((SpO2_i-SaO2_i )^2 ))/n.
Time Frame: 1-5 hours
Measure: Number; unit: % of oxygen saturated hemoglobin
Arm/Group | MightySat
Number analyzed (Participants) | 39
% of oxygen saturated hemoglobin | 1.30

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | MightySat
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 13/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MightySat (N=39)
Anxiety (Nervous system disorders) | 1
Dizziness/Lightheadedness (Nervous system disorders) | 3
Arterial line (healing) (Surgical and medical procedures) | 3
Hypotension (Cardiac disorders) | 2
Abnormal ECG (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT05083351/Prot_SAP_001.pdf